CLINICAL TRIAL: NCT06863584
Title: A Phase II Trial of Stereotactic Body Radiotherapy (SBRT) With Lenalidomide Maintenance for Solitary Plasmacytoma
Brief Title: SBRT Plus Lenalidomide for Solitary Plasmacytoma: Phase II Trial
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Y2025-0115
Record Dates: First submitted 2025-03-03; First posted 2025-03-07 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-02

CONDITIONS: Solitary Plasmacytoma
Keywords: sbrt; solitary plasmacytoma; Lenalidomide
MeSH Terms: conditions — Neoplasms, Plasma Cell | interventions — Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- SBRT Plus Lenalidomide (Experimental): The SBRT will deliver a dose of 30Gy in 5 fractions to the planning target volume (PTV) and/or 35Gy in 5 fractions to the planning gross tumor volume (PGTV). The specific regimen will be determined based on patient's medical condition and tumor characteristics. Lenalidomide will be taken orally at a dose of 10mg, starting from the first day after the completion of radiotherapy, for 21 consecutive days, followed by a 7-day rest period. This cycle will be repeated for a total of four cycles.
  Interventions: Drug: Lenalidomide (Revlimid); Radiation: SBRT

INTERVENTIONS:
Drug: Lenalidomide (Revlimid) — 10mg po for 21 days, followed by a 7-day rest period.
Radiation: SBRT — PTV 30Gy/5f and/or PGTV 35Gy/5F.

SUMMARY:
Solitary Plasmacytoma (SP) is a rare malignant plasma cell tumor, including Solitary Bone Plasmacytoma (SBP) and Solitary Extramedullary Plasmacytoma (SEP). Radiotherapy is the preferred treatment for SP. Although the local response rate of SP after radiotherapy is as high as 86%, 55% of patients will experience disease progression within 5 years.

Stereotactic Body Radiation Therapy (SBRT), as a new technology for "precision radiotherapy," delivers a higher dose of radiation to the tumor site through a few short treatment sessions while maintaining low-dose exposure to surrounding normal tissues. This approach achieves good local tumor control and effectively reduces radiotherapy-related side effects, making it valuable for application in SP patients. Additionally, numerous preclinical studies have confirmed that SBRT has positive immunomodulatory effects.

Based on data published in the New England Journal of Medicine in 2013, lenalidomide-based immunomodulatory therapy significantly delays the progression of symptomatic myeloma with minimal toxicity in patients with smoldering multiple myeloma.

This study aims to assess the efficacy and safety of combining SBRT with lenalidomide in patients with SP, compared to conventional intensity-modulated radiotherapy. The goal is to extend progression-free survival (PFS) in newly diagnosed SP patients, reduce adverse reactions, and improve quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Patients with newly diagnosed solitary plasmacytoma (SP).
* Age between 18 and 80 years.
* Diagnosis of SP must meet the following four criteria:

Biopsy-confirmed plasmacytoma in bone or soft tissue. No evidence of clonal plasma cell proliferation in the bone marrow. No other lesions detected on whole-body imaging (whole-body PET-CT or MRI recommended) except for the primary solitary lesion.

No end-organ damage caused by plasma cell disease, including SLiM CRAB [excluding bone destruction caused by the SP itself.

Exclusion Criteria:

* Patients who are not suitable for radiotherapy or unable to receive SBRT due to technical limitations, such as patients with plasmacytoma in the extremities who cannot abduct the affected limb or maintain the treatment position due to pain.
* Eastern Cooperative Oncology Group (ECOG) performance status score greater than 2.
* Patients who meet the diagnostic criteria for multiple myeloma at the time of diagnosis: bone marrow biopsy showing more than 10% plasma cells, serum calcium level above 11.5 mg/dL, serum creatinine above 2 mg/dL, creatinine clearance rate below 40 mL/min, or hemoglobin below 10 g/dL.
* Patients with uncontrolled infectious comorbidities.
* Patients with other active malignancies.
* Pregnant or breastfeeding patients.
* Patients with a history or current pulmonary embolism.
* Patients with a history of autoimmune disease, even if it is controlled.
* Patients who are seropositive for human immunodeficiency virus (HIV), hepatitis C virus (HCV), or hepatitis B virus (HBV) DNA > 1,000 copies/mL.
* Patients with myocardial infarction within 6 months prior to enrollment, New York Heart Association (NYHA) Class III or IV heart failure, uncontrolled angina, or severe uncontrolled arrhythmia.
* Patients with neuropathy Grade 2 or higher according to the National Cancer Institute Common Terminology Criteria for Adverse Events.
* Patients with neutrophil count < 1×10^9/L, hemoglobin < 8 g/dL, or platelet count < 75×10^9/L.
* Patients with severely impaired liver or kidney function: alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > 3 × upper limit of normal (ULN), total bilirubin > 1.5 × ULN, or estimated glomerular filtration rate (eGFR) < 40 mL/min.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Estimated)
Dates: Start 2025-02-10 (Actual); Primary Completion 2027-03-31 (Estimated); Study Completion 2032-03-01 (Estimated)

PRIMARY OUTCOMES:
PFS | 5 years
  PFS measures the percentage of patients who remain free from disease progression over a five-year period.

SECONDARY OUTCOMES:
OS | 5 years
  OS was calculated from the enrollment to death

CONTACTS AND LOCATIONS:
Locations (1):
- 2nd Affiliated Hospital, School of Medicine, Hangzhou, Zhejiang, China